CLINICAL TRIAL: NCT00945737
Title: A Randomized, Controlled Parallel Study to Evaluate the Effects of a Non-Commercial Soy Protein Product on Fecal Bile Acids and Blood Lipids in Men and Women With Mild to Moderate Hypercholesterolemia
Brief Title: A Study on the Effects of Soy Protein on Blood Lipids in Men and Women With Mild to Moderate Hypercholesterolemia
Acronym: PRV-08009
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solae, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRV-08009
Record Dates: First submitted 2009-07-21; First posted 2009-07-24 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; cholesterol; soy
MeSH Terms: conditions — Hypercholesterolemia | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy protein (Active Comparator)
  Interventions: Dietary Supplement: Soy protein; 25 grams/day
- Milk protein (Placebo Comparator)
  Interventions: Dietary Supplement: Control protein

INTERVENTIONS:
Dietary Supplement: Soy protein; 25 grams/day — Soy protein
  Arms: Soy protein
Dietary Supplement: Control protein — Milk protein
  Arms: Milk protein

SUMMARY:
The objectives of the trial are to determine whether a non-commercial soy protein product, consumed as part of a low-saturated fat diet, reduces low-density lipoprotein cholesterol (LDL-C) concentrations in men and women with mild to moderate hypercholesterolemia, and affects other aspects related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-79 years of age
* Fasting LDL-Cholesterol level borderline to high range taking no cholesterol lowering medications
* otherwise judged to be in good health, willing to maintain a stable body weight and follow the TLC diet throughout the trial.

Exclusion Criteria:

* CHD or CHD risk equivalent
* Pregnancy
* Food allergy or sensitivity to soy or milk protein
* Certain muscle, liver, kidney, lung or gastrointestinal conditions and medications
* Poorly controlled hypertension
* Cancer treated within prior 2 years

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The difference between treatment groups in the percent change from baseline to the end of treatment in LDL-C | 4 weeks

SECONDARY OUTCOMES:
Changes in other lipid levels and other related biomarkers | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Reeves, DO, Principal Investigator — Provident Clinical Research; Mano Patri, MD, Principal Investigator — Provident Clinical Research, Addison, IL
Locations (2):
- United States (2):
  - Provident Clinical Research, Addison, Illinois
  - Provident Clinical Research, Bloomington, Indiana

REFERENCES:
- [Derived] Maki KC, Butteiger DN, Rains TM, Lawless A, Reeves MS, Schasteen C, Krul ES. Effects of soy protein on lipoprotein lipids and fecal bile acid excretion in men and women with moderate hypercholesterolemia. J Clin Lipidol. 2010 Nov-Dec;4(6):531-42. doi: 10.1016/j.jacl.2010.09.001. Epub 2010 Oct 1. PMID 21122701